CLINICAL TRIAL: NCT05649358
Title: Pilot Testing a Novel Non-invasive Lactate Sensor Using Split Ring Low Energy Microwave Sensors
Brief Title: Pilot Testing a Novel Non-invasive Lactate Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00115293
Record Dates: First submitted 2022-08-18; First posted 2022-12-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-06

CONDITIONS: Hyperlactatemia
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Intervention Model Description: The investigators will test the device on 8 male and 8 female participants to determine if there are any sex differences in the performance of the sensor. As there is likely going to be inter-individual variability in the participants, the investigators have chosen to test 8 males and 8 females rather than 5 and 5 as suggested by the reviewer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of non-invasive lactate sensor (Experimental): To determine the efficacy and accuracy of the non-invasive lactate sensor
  Interventions: Device: Lactate sensor (Lactisense)

INTERVENTIONS:
Device: Lactate sensor (Lactisense) — Non-invasive monitoring of interstitial lactate levels during and after exercise.

SUMMARY:
To test the efficacy and accuracy of a novel non-invasive lactate sensor in humans undergoing strenuous leg exercise.

DETAILED DESCRIPTION:
The study investigators have designed a novel non-invasive lactate sensor (Lactisense) Lactisense is a planar, flexible, passive, chip-less resonator that can be taped to the skin in order to measure lactate levels in the body. It sends a signal to a nearby reader, which can be translated into a concentration value. It has so far been tested in the lab with good accuracy, but has not been tested on humans. The sensors are designed to use very low energy microwaves that can detect alterations in interstitial and muscle metabolites.

In this study the investigators will test the sensor by having participants perform strenuous exercise (lifting weights) with Lactisense sensors attached to their skin on the top of the thigh and upper arm to evaluate lactate levels at the site of production and systemic levels respectively. The exercise will be performed using a well-established protocol to elevate lactate levels using a leg-press weights machine. The investigators will use a commercial capillary blood lactate meter (via finger prick) to verify whether lactate levels are actually changing in the body, and use Lactisense to try to measure these changes and compare to the values obtained using the commercial capillary blood lactate meter.

ELIGIBILITY:
Inclusion Criteria:

Healthy and physically active volunteers

Exclusion Criteria:

Existing health conditions e.g blood pressure > 150/95, joint injury that would contraindicate exercise. Individuals who answer "yes" to any of the health condition questions on the PAR-Q questionnaire will also be excluded. As ketones might interfere with the sensor signal, we will exclude anyone with metabolic conditions or following a ketogenic diet.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
That the lactate sensor under test is able track increase in interstitial lactate levels in exercising humans that follow the same time course as lactate values obtained from a commercial blood capillary lactate monitor. | 6 months
  The novel sensor data will be compared to lactate values measured simultaneously with a commercial blood capillary lactate monitor in exercising humans.

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Light, PhD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Diabetes Institute, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No